CLINICAL TRIAL: NCT02088918
Title: A Open-label, Single-dose, 2-Sequence, 2-Period, Crossover Study to Assess Safety and Pharmacokinetics of a Nateglinide/Metformin HCl Combined Tablet Compared With a Nateglinide 120 mg Tablet and Metformin HCl 500 mg Tablet Under Fasting Conditions in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID_Fasticmet_1201
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Nateglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nateglinide+Metformin (Active Comparator): coadministration of nateglinide and metformin
  Interventions: Drug: Nateglinide; Drug: Metformin
- Nateglinide/Metformin (Experimental): Nateglinide/Metformin tablet
  Interventions: Drug: Nateglinide/Metformin

INTERVENTIONS:
Drug: Nateglinide
  Arms: Nateglinide+Metformin
Drug: Nateglinide/Metformin
  Arms: Nateglinide/Metformin
Drug: Metformin
  Arms: Nateglinide+Metformin

SUMMARY:
A Randomized, Open-label, Single-dose, 2-Sequence, 2-Period, Crossover Study to Assess Safety and Pharmacokinetics of a Nateglinide/Metformin HCl Combined Tablet Compared with a Nateglinide 120 mg Tablet and Metformin HCl 500 mg Tablet under Fasting Conditions in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 40
* Signed informed consent

Exclusion Criteria:

* Has a history of hypersensitivity to IP ingredients
* Hypertension or hyportension

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
AUC last | 0-~24hrs
Cmax | 0~24hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam University Hospital, Daejeon, South Korea